CLINICAL TRIAL: NCT05243004
Title: Assessment of a Phone Nurse Consultation Benefit on Compliance With the PreOperative Instructions for Patients Undergoing Scheduled Surgery and Entering the Operation Day
Brief Title: Phone Nurse Consultation Benefit on Compliance With PreOperative Instructions for Patients Undergoing Scheduled Surgery
Acronym: CIT-PO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021_0069
Record Dates: First submitted 2022-02-03; First posted 2022-02-16 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Nurse Consultation (Experimental): Patients will benefit, in addition to the usual care, including a reminder by the secretary of the PORU the day before the operation, a phone call from nurse no later than 72 hours before surgery to explain and remind them of the instructions for preoperative preparation and answer any questions they may have.
  Interventions: Other: Phone Nurse consultation
- Standard care (No Intervention): Patients in this group will follow the usual preparation schedule including a reminder by the secretary of the PORU the day before the operation.

INTERVENTIONS:
Other: Phone Nurse consultation — A phone call will be made by the nurse 72 hours before the surgery. During this phone call, the nurse :
  * underlines the preoperative preparation instructions (skin preparation, fasting period, specific medical instructions given by the anesthesiologist, administrative instructions)
  * ensures that the reason for hospitalization is understood
  * answers the patient's questions.
  Arms: Phone Nurse Consultation

SUMMARY:
A preoperative reception unit (PORU) has been created at Foch Hospital to receive patients needing surgery and entering the same day of the operation (D0) as part of the reduction in average lengths of stay. This new mode of care requires a specific organization which requires the patient to become the main actor in his preparation.To optimize and make this new care fluid, a phone nurse consultation has been set up to support patients. The objective of this consultation is to discuss with the patient the different stages of his journey. The nurse checks the patient's level of information and reformulates if necessary so that he can receive clear and appropriate information, verifies that the patient has correctly integrated all that is expected for his preoperative preparation. It thus makes it possible to anticipate the issues that could impact the patient care process.The relevance of this consultation has never been assessed. However, the nurses have always good feedback from patients who are often surprised, satisfied with this interview and attentive. On the other hand, nurses who receive patients on the day of their intervention in PORU observe better fluidity in the care of patients who have had a phone nurse consultation. The patient is better prepared, which allows simpler and faster care.

This randomized controlled study will allow investigators to validate the perception of nurse and to assess the relevance of this phone nurse consultation in the best preoperative preparation of patients, the management of preoperative anxiety and the fluidity of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or over,
* Willing to undergo a scheduled surgery at Foch Hospital and entering the hospital the same morning of his intervention in the Preoperative Reception Unit (PORU),
* Having a scheduled pre-anesthetic consultation visit,
* Having signed a consent form,
* Affiliated with a health insurance plan.

Exclusion Criteria:

* Patient who does not speak or understand French,
* Patient requiring an invasive radiology procedure,
* Patient deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Compliance with preoperative medical preparation instructions between the 2 groups (with and without preoperative nurse consultation). | At the intervention day (just before surgery)
  The preoperative medical preparation will be assessed by a composite criterion including compliance with:
  * skin preparation (shower and depilation if applicable)
  * preoperative fasting
  * medical instructions (stopping or continuing drug treatments)

SECONDARY OUTCOMES:
Compliance with preoperative administrative preparation instructions between the 2 groups (with and without preoperative telephone nurse consultation). | At the intervention day (just before surgery)
  The preoperative administrative preparation will be assessed by the following 2 criteria:
  * the time of arrival,
  * instructions for filling in administrative documents (care consent, person to be notified, trustworthy, etc.).
Benefit of a preoperative nurse consultation on patient anxiety | at inclusion and at the intervention day (just before surgery)
  Anxiety will be assessed using a numerical scale from 0 (no anxiety) to 10 (highest level of anxiety)
Patient's satisfaction regarding preoperative support | At the intervention day (just before surgery)
  Satisfaction will be assessed using the patient support satisfaction assessment questionnaire (from "Not at all satisfied" to "Very satisfied")
Patient's satisfaction regarding the phone nurse consultation | At the intervention day (just before surgery)
  Satisfaction will be assessed using the satisfaction assessment questionnaire for the phone nurse consultation (from "Useless" to "Essential"

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Hullier-Ammar, Principal Investigator — Foch Hospital
Locations (1):
- Foch Hospital, Suresnes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No